CLINICAL TRIAL: NCT03738241
Title: A Phase II Study to Assess the Safety, Reactogenicity and Immunogenicity of a Single Dose of 2017 A/H7N9 Inactivated Influenza Vaccine (IIV) Administered Intramuscularly With or Without AS03 Adjuvant in 2013 A/H7N9 IIV Primed or A/H7 IIV Naïve Subjects
Brief Title: 2017 A/H7N9 IIV Revaccination
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 17-0090; HHSN272201300015I
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2021-07-01 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2018-11-08

CONDITIONS: Avian Influenza; Influenza Immunisation
Keywords: A/H7N9 Inactivated Influenza Vaccine; AS03 Adjuvant; Immunogenicity; Influenza; Phase II; Reactogenicity; Safety; Vaccine
MeSH Terms: conditions — Influenza in Birds; Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Arm 1 (Experimental): Participants will have prior administration of 2013 A/H7N9 IIV with MF59. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 (n=50) or 3.75 mcg HA per 0.5 ml dose of 2017 A/H7N9 IIV unadjuvanted administered intramuscularly on Day 1 (n=50). Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 2 (Experimental): Participants will have prior administration of 2013 A/H7N9 IIV with AS03. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 (n=50) or 3.75 mcg HA per 0.5 ml dose of 2017 A/H7N9 IIV unadjuvanted administered intramuscularly on Day 1 (n=50). Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 3 (Experimental): Participants will have prior administration of 2013 A/H7N9 IIV 15 mcg or 45 mcg unadjuvanted. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 (n=50) or 3.75 mcg HA per 0.5 ml dose of 2017 A/H7N9 IIV unadjuvanted administered intramuscularly on Day 1 (n=50). Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 4 (Experimental): Participants will have prior administration of 2013 A/H7N9 IIV + MF59 or AS03 (1st) then 2013 A/H7N9 IIV 15 mcg (2nd). Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 (n=30) or 3.75 mcg HA per 0.5 ml dose of 2017 A/H7N9 IIV unadjuvanted administered intramuscularly on Day 1 (n=30). Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent
- Arm 5 (Experimental): Participants who are A/H7 IIV-Naïve. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1 (n=30) or 3.75 mcg HA per 0.5 ml dose of 2017 A/H7N9 IIV unadjuvanted administered intramuscularly on Day 1 (n=30). Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Interventions: Biological: A/H7N9; Drug: AS03; Other: Phosphate Buffered Saline (PBS) diluent

INTERVENTIONS:
Biological: A/H7N9 — Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and the PB2, PB1, PA, NP, M and NS from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
Drug: AS03 — AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
Other: Phosphate Buffered Saline (PBS) diluent — 0.006M PBS diluent for Influenza Virus Vaccine.

SUMMARY:
This is a Phase II clinical trial in up to 420 males and non-pregnant females, 19 to 70 years of age, inclusive, who are in good health and meet all eligibility criteria. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of one dose of a monovalent inactivated split influenza 2017 A/H7N9 virus vaccine (2017 A/H7N9 IIV), administered intramuscularly (IM) at 3.75 mcg hemagglutinin (HA) per dose, given with or without AS03 adjuvant to subjects primed with a monovalent inactivated split influenza 2013 A/H7N9 virus vaccine (2013 A/H7N9 IIV) in DMID Protocols 13-0032 and 13-0033, or to those who are A/H7 IIV-naïve. Phosphate buffered saline (PBS) diluent will be used to achieve the targeted dosage. The study will be conducted at 9 Vaccine and Treatment Evaluation Unit (VTEU) sites (including their subcontractors). Study duration is approximately 17 months with subject participation duration up to 13 months. The primary objectives are: 1) to assess the safety and reactogenicity of 2017 A/H7N9 IIV given with or without AS03 adjuvant following receipt of one dose of study vaccine; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of the study vaccine.

DETAILED DESCRIPTION:
This is a Phase II clinical trial in up to 420 males and non-pregnant females, 19 to 70 years of age, inclusive, who are in good health and meet all eligibility criteria, which include a screening erythrocyte sedimentation rate (ESR) laboratory evaluation. This clinical trial is designed to assess the safety, reactogenicity and immunogenicity of one dose of a monovalent inactivated split influenza 2017 A/H7N9 virus vaccine (2017 A/H7N9 IIV) manufactured by Sanofi Pasteur (SP), administered intramuscularly (IM) at 3.75 mcg hemagglutinin (HA) per dose, given with or without AS03 adjuvant manufactured by GlaxoSmithKline Biologicals (GSK), to subjects primed with a monovalent inactivated split influenza 2013 A/H7N9 virus vaccine (2013 A/H7N9 IIV) in DMID Protocols 13-0032 and 13-0033, or to those who are A/H7 IIV-naïve. Phosphate buffered saline (PBS) diluent manufactured by Patheon Manufacturing Services LLC will be used to achieve the targeted dosage. Subjects who received the 2013 A/H7N9 IIV in DMID Protocols 13-0032 and 13-0033 or are A/H7 IIV-naïve will be stratified by prior receipt of 2013 A/H7N9 IIV, as well as by site and prior receipt of licensed, seasonal influenza vaccine (defined as receipt of at least one of the 2017-2018 and/or 2018-2019 licensed, seasonal influenza vaccines versus none), then randomly assigned in a 1:1 ratio to 1 of 2 treatment arms to receive 1 dose of 2017 A/H7N9 IIV at 3.75 mcg HA per dose with or without AS03 adjuvant. The study will be conducted at 9 Vaccine and Treatment Evaluation Unit (VTEU) sites (including their subcontractors). Study duration is approximately 17 months with subject participation duration up to 13 months. The primary objectives are: 1) to assess the safety and reactogenicity of 2017 A/H7N9 IIV given with or without AS03 adjuvant following receipt of one dose of study vaccine; 2) to assess the serum hemagglutination inhibition (HAI) and neutralizing (Neut) antibody responses following receipt of the study vaccine. Secondary objectives are: 1) to assess unsolicited non-serious adverse events (AEs) following receipt of the study vaccine; 2) to assess medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs), following receipt of the study vaccine; 3) To assess the kinetics and durability of serum HAI and Neut antibody responses following receipt of the study vaccine.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible to participate in this trial must meet all of the following inclusion criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Must agree to the collection of venous blood per protocol.
4. Must agree to have residual specimens and samples/specimens collected during this trial specifically for the purpose of future research stored for future research use.
5. Are males or non-pregnant females, 19 to 70 years of age, inclusive.
6. Are in good health* *As determined by medical history and physical examination to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, which would affect the assessment of the safety of subjects or the immunogenicity of study vaccinations. Chronic medical diagnoses or conditions should be stable for the last 60 days (no hospitalizations, emergency room or urgent care for condition and no adverse symptoms that need medical intervention such as medication change/supplemental oxygen). This includes no change in chronic prescription medication, dose or frequency as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site PI or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site PI or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to study vaccination. Note: Topical, nasal and inhaled medications (except inhaled corticosteroids as outlined in the Subject Exclusion Criteria as well as herbals, vitamins and supplements are permitted.
7. Oral temperature is less than 100.0 degrees Fahrenheit.
8. Pulse is 47 to 100 beats per minute, inclusive.
9. Systolic blood pressure is 85 to 150 mmHg, inclusive.
10. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
11. Erythrocyte Sedimentation Rate (ESR) is less than 30 mm per hour.
12. Women of childbearing potential** must use an acceptable contraception method*** from 30 days before study vaccination until 60 days after study vaccination.

    **Not sterilized via tubal ligation, bilateral oophorectomy, salpingectomy, hysterectomy, or successful Essure(R) placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year has passed since the last menses if menopausal.

    ***Includes non-male sexual relationships, abstinence from sexual intercourse with a male partner, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the study vaccination, barrier methods such as condoms or diaphragms/cervical cap with spermicide, effective intrauterine devices, NuvaRing(R), and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
13. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to study vaccination.
14. Received 1 or 2 doses of 2013 A/H7N9 IIV with or without AS03 or MF59 adjuvant in DMID Protocols 13-0032 or 13-0033, or are A/H7 IIV-naïve.

Exclusion Criteria:

Subjects eligible to participate in this trial must not meet any of the following exclusion criteria:

1. Have an acute illness*, as determined by the site PI or appropriate sub-investigator, within 72 hours prior to study vaccination.

   *An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site PI or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site PI or appropriate sub-investigator, is a contraindication to study participation**.

   **Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this trial.
3. Have immunosuppression as a result of an underlying illness or treatment, a recent history or current use of immunosuppressive or immunomodulating disease therapy.
4. Use of cytotoxic anticancer chemotherapy or radiation therapy within 3 years prior to study vaccination.
5. Have known active neoplastic disease or a history of any hematologic malignancy. Non-melanoma, treated, skin cancers are permitted.
6. Have known human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection.
7. Have known hypersensitivity or allergy to eggs, egg or chicken protein, squalene-based adjuvants, or other components of the study vaccine.
8. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza vaccines.
9. Have a personal or family history of narcolepsy.
10. Have a history of Guillain-Barré Syndrome (GBS).
11. Have a history of convulsions or encephalomyelitis within 90 days prior to study vaccination.
12. Have a history of Potentially Immune-Mediated Medical Conditions (PIMMCs).
13. Have a history of alcohol or drug abuse within 5 years prior to study vaccination.
14. Have any diagnosis, current or past, of schizophrenia, bipolar disease or other psychiatric diagnosis that may interfere*** with subject compliance or safety evaluations.

    ***As determined by the site PI or appropriate sub-investigator.
15. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to study vaccination.
16. Have taken oral or parenteral (including intra-articular) corticosteroids of any dose within 30 days prior to study vaccination.
17. Have taken high-dose inhaled corticosteroids**** within 30 days prior to study vaccination.

    ****High-dose defined as per age as using inhaled high-dose per reference chart in the National Heart, Lung and Blood Institute Guidelines for the Diagnosis and Management of Asthma (EPR-3) or other lists published in UPTODATE.
18. Received or plan to receive a licensed, live vaccine within 30 days before or after study vaccination.
19. Received or plan to receive a licensed, inactivated vaccine (excluding all licensed, seasonal IIVs) within 14 days before or after study vaccination.
20. Received or plan to receive a licensed, seasonal IIV within 21 days before or after study vaccination.
21. Received immunoglobulin or other blood products (except Rho D immunoglobulin) within 90 days prior to study vaccination.
22. Received an experimental agent***** within 30 days prior to study vaccination or expect to receive an experimental agent****** during the trial-reporting period*******.

    *****Including vaccine, drug, biologic, device, blood product, or medication.

    ******Other than from participation in this trial.

    *******Approximately 12 months after study vaccination.
23. Are participating or plan to participate in another clinical trial with an interventional agent******** that will be received during the trial-reporting period*********.

    ********Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.

    *********Approximately 12 months after study vaccination.
24. Have a history of influenza A/H7 subtype infection.
25. Had substantial direct contact********** with live or freshly slaughtered poultry or pigeons while in mainland China within the past five years.

    **********Substantial direct contact is defined as visited a poultry farm and/or a live poultry market.
26. Occupational exposure to or substantial direct physical contact*********** with birds in the past year and through 21 days after study vaccination.

    ***********Exposure to free range chickens in the yard is exclusionary. Casual contact with birds at petting zoos or county or state fairs or having pet birds does not exclude subjects from study participation.
27. Female subjects who are breastfeeding.
28. Plan to travel outside the US (continental US, Hawaii and Alaska) from the time of study vaccination through 21 days after study vaccination.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-06-19 (Actual); Study Completion 2020-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Emory Children's Center - Pediatric Infectious Diseases, Atlanta, Georgia
  - University of Iowa - Vaccine Research and Education Unit, Iowa City, Iowa
  - University of Maryland Baltimore - School of Medicine - Medicine, Baltimore, Maryland
  - Saint Louis University - Center for Vaccine Development, St Louis, Missouri
  - Cincinnati Children's Hospital Medical Center - Infectious Diseases, Cincinnati, Ohio
  - Vanderbilt University Medical Center - Infectious Diseases, Nashville, Tennessee
  - The University of Texas Medical Branch - Sealy Center for Vaccine Development (SCVD), Galveston, Texas
  - Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas
  - Kaiser Permanente Washington Health Research Institute - Vaccines and Infectious Diseases, Seattle, Washington

REFERENCES:
- [Derived] El Sahly HM, Anderson EJ, Jackson LA, Neuzil KM, Atmar RL, Bernstein DI, Chen WH, Creech CB, Frey SE, Goepfert P, Meier J, Phadke V, Rouphael N, Rupp R, Stapleton JT, Spearman P, Walter EB, Winokur PL, Yildirim I, Williams TL, Oshinsky J, Coughlan L, Nijhuis H, Pasetti MF, Krammer F, Stadlbauer D, Nachbagauer R, Tsong R, Wegel A, Roberts PC. Anti-neuraminidase and anti-hemagglutinin stalk responses to different influenza a(H7N9) vaccine regimens. Vaccine. 2025 Feb 15;47:126689. doi: 10.1016/j.vaccine.2024.126689. Epub 2025 Jan 4. PMID 39756216
- [Derived] El Sahly HM, Yildirim I, Frey SE, Winokur P, Jackson LA, Bernstein DI, Creech CB, Chen WH, Rupp RE, Whitaker JA, Phadke V, Hoft DF, Ince D, Brady RC, Edwards KM, Ortiz JR, Berman MA, Weiss J, Wegel A; DMID 17-0090 Study Group. Safety and Immunogenicity of a Delayed Heterologous Avian Influenza A(H7N9) Vaccine Boost Following Different Priming Regimens: A Randomized Clinical Trial. J Infect Dis. 2024 Feb 14;229(2):327-340. doi: 10.1093/infdis/jiad276. PMID 37466221

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were healthy males and non-pregnant females between 19 and 70 years old, inclusively. They were recruited from the communities at large around the clinical sites. Participants were enrolled between 18DEC2018 and 19MAR2019.
Groups:
- 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV: Participants will have prior administration of 2013 A/H7N9 IIV with MF59. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03: Participants will have prior administration of 2013 A/H7N9 IIV with MF59. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Drug: AS03 AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV: Participants will have prior administration of 2013 A/H7N9 IIV with AS03. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03: Participants will have prior administration of 2013 A/H7N9 IIV with AS03. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Drug: AS03 AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV|2017 A/H7N9 IIV: Participants will have prior administration of 2013 A/H7N9 IIV 15 mcg or 45 mcg unadjuvanted. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03: Participants will have prior administration of 2013 A/H7N9 IIV 15 mcg or 45 mcg unadjuvanted. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Drug: AS03 AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV: Participants will have prior administration of 2013 A/H7N9 IIV + MF59 or AS03 (1st) then 2013 A/H7N9 IIV 15 mcg (2nd). Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03: Participants will have prior administration of 2013 A/H7N9 IIV + MF59 or AS03 (1st) then 2013 A/H7N9 IIV 15 mcg (2nd). Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Drug: AS03 AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- A/H7 IIV Naïve |2017 A/H7N9 IIV: Participants who are A/H7 IIV-Naïve. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
- A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03: Participants who are A/H7 IIV-Naïve. Then, 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1. Phosphate buffered saline (PBS) diluent may be used to achieve targeted dosages.
  Biological: A/H7N9 Monovalent split 2017 A/H7N9 Inactivated Influenza Virus Vaccine containing the Hemagglutinin (HA) and Neuraminidase (NA) from low pathogenic avian influenza A/Hong Kong/125/2017 (H7N9) and other components from A/Puerto Rico/8/1934 (H1N1). The HA content of the 2017 A/H7N9 vaccine formulations were determined by Single Radial Immunodiffusion (SRID) assay to be approximately two times higher (14.45 mcg of HA per 0.5 mL dose) than the targeted HA content on the label (7.5 mcg of HA per 0.5 mL dose).
  Drug: AS03 AS03 oil-in-water emulsion-based adjuvant system containing DL-alpha-tocopherol, squalene, polysorbate 80, and a buffer.
  Other: Phosphate Buffered Saline (PBS) diluent 0.006M PBS diluent for Influenza Virus Vaccine.
Period: Overall Study
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Started | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Completed | 37 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 34
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants
Groups:
- 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV: 2013 A/H7N9 IIV with MF59. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03: 2013 A/H7N9 IIV with MF59. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV: 2013 A/H7N9 IIV with AS03. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03: 2013 A/H7N9 IIV with AS03. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV|2017 A/H7N9 IIV: 2013 A/H7N9 IIV 15 mcg or 45 mcg unadjuvanted. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03: 2013 A/H7N9 IIV 15 mcg or 45 mcg unadjuvanted. 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV: 2013 A/H7N9 IIV + MF59 or AS03 (1st) then 2013 A/H7N9 IIV 15 mcg (2nd). 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1.
- 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03: 2013 A/H7N9 IIV + MF59 or AS03 (1st) then 2013 A/H7N9 IIV 15 mcg (2nd). 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1.
- A/H7 IIV Naïve |2017 A/H7N9 IIV: 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) unadjuvanted administered intramuscularly on Day 1.
- A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03: 3.75 mcg Hemagglutinin (HA) per 0.5 ml dose of 2017 A/H7N9 Inactivated Influenza Virus Vaccine (IIV) + AS03 adjuvant administered intramuscularly on Day 1.
- Total: Total of all reporting groups
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03 | Total
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35 | 304
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 19 - 35 years | 9 | 4 | 5 | 1 | 11 | 5 | 5 | 4 | 20 | 19 | 83
  Age, Categorical: 36 - 50 years | 14 | 18 | 6 | 6 | 11 | 15 | 3 | 3 | 3 | 10 | 89
  Age, Categorical: 51-70 years | 15 | 18 | 13 | 11 | 18 | 24 | 12 | 9 | 6 | 6 | 132
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 11 | 16 | 26 | 25 | 11 | 13 | 16 | 15 | 172
  Male | 20 | 19 | 13 | 2 | 14 | 19 | 9 | 3 | 13 | 20 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3 | 0 | 2 | 3 | 0 | 2 | 4 | 4 | 21
  Not Hispanic or Latino | 37 | 38 | 21 | 18 | 38 | 41 | 20 | 14 | 25 | 31 | 283
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Asian | 0 | 1 | 1 | 0 | 1 | 2 | 1 | 1 | 4 | 2 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 3 | 1 | 2 | 2 | 4 | 0 | 3 | 10 | 11 | 42
  White | 30 | 35 | 22 | 13 | 34 | 34 | 18 | 11 | 12 | 20 | 229
  More than one race | 2 | 1 | 0 | 2 | 2 | 4 | 1 | 0 | 3 | 1 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35 | 304
Body Mass Index (BMI) [Count of Participants; unit: Participants]
  < 30 kg/m^2 | 25 | 26 | 16 | 13 | 29 | 28 | 15 | 8 | 17 | 26 | 203
  >= 30 kg/m^2 | 13 | 14 | 8 | 5 | 11 | 16 | 5 | 8 | 12 | 9 | 101
Prior Seasonal Influenza Vaccination [Count of Participants; unit: Participants]
  2017-2018 and 2018-2019 | 30 | 32 | 17 | 13 | 31 | 30 | 16 | 10 | 13 | 14 | 206
  2017-2018 only | 0 | 2 | 3 | 1 | 2 | 2 | 1 | 2 | 6 | 7 | 26
  2018-2019 only | 3 | 3 | 0 | 1 | 2 | 6 | 0 | 3 | 4 | 6 | 28
  Neither | 5 | 3 | 4 | 3 | 5 | 6 | 3 | 1 | 6 | 8 | 44

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies on Day 22 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: The modified intent-to-treat (mITT) population includes all participants who received study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 22.7 [14.5 to 35.8] | 116.1 [82.1 to 164.2] | 77.7 [44.7 to 135.1] | 190.3 [100.9 to 358.9] | 10.9 [7.5 to 15.9] | 31.7 [21.3 to 47.0] | 33.1 [17.0 to 64.1] | 180.9 [100.5 to 325.7] | 6.6 [4.9 to 8.9] | 8.3 [6.0 to 11.5]

2. Primary Outcome: Geometric Mean Titers (GMT) of Serum Neutralizing (Neut) Antibodies on Day 22 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: The modified intent-to-treat (mITT) population includes all participants who received study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for Neut antibody assays for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 64.3 [39.3 to 105.2] | 367.6 [251.9 to 536.4] | 204.5 [112.6 to 371.6] | 870.9 [623.7 to 1216.0] | 28.6 [17.8 to 46.1] | 72.2 [47.3 to 110.2] | 115.1 [54.0 to 245.2] | 562.0 [316.0 to 999.4] | 5.8 [4.9 to 6.9] | 10.8 [7.7 to 15.1]

3. Primary Outcome: Number of Participants Reporting Serious Adverse Events (SAEs)
Description: SAEs included any untoward medical occurrence that resulted in death; was life threatening; was a persistent/significant disability/incapacity; required inpatient hospitalization or prolongation or a congenital anomaly/birth defect.
Time Frame: Day 1 through Day 366
Population: The safety population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

4. Primary Outcome: Number of Participants Reporting Clinical Safety Laboratory Adverse Events (AEs)
Description: Laboratory parameters include alanine aminotransferase (ALT), bilirubin, creatinine, hemoglobin, platelets and white blood cells (WBC). Thresholds for adverse events were considered as ALT 44 IU/L or greater (female) or 61 IU/L or greater (male); bilirubin 1.30 mg/dL or greater; creatinine 1.1 mg/dL or greater (female) or 1.4 mg/dL or greater (male); hemoglobin 11.4 g/dL or lower (female) or 12.4 g/dL or lower (male); platelets 139 x10^3/µL or below or 416 x10^3/µL or greater; or WBC or 3.9 x10^3/µL or lower or 10.6 x10^3/µL or higher.
Time Frame: Day 1 to Day 8
Population: The safety population includes all participants who received study vaccination. Participants with at least one lab result reported for Day 8 were included for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants
  ALT: number analyzed (Participants) | 37 | 40 | 24 | 18 | 40 | 43 | 20 | 16 | 28 | 34
  ALT | 1 | 0 | 3 | 0 | 3 | 0 | 1 | 3 | 0 | 1
  Bilirubin: number analyzed (Participants) | 37 | 40 | 24 | 18 | 40 | 43 | 20 | 16 | 28 | 34
  Bilirubin | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine: number analyzed (Participants) | 37 | 40 | 24 | 18 | 40 | 43 | 20 | 16 | 28 | 34
  Creatinine | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1
  Hemoglobin: number analyzed (Participants) | 37 | 40 | 24 | 17 | 39 | 41 | 20 | 16 | 28 | 35
  Hemoglobin | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 1 | 3
  Platelets: number analyzed (Participants) | 37 | 40 | 24 | 17 | 39 | 41 | 20 | 16 | 28 | 35
  Platelets | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  WBC: number analyzed (Participants) | 37 | 40 | 24 | 17 | 39 | 41 | 20 | 16 | 28 | 35
  WBC | 3 | 2 | 2 | 0 | 3 | 3 | 0 | 1 | 1 | 3

5. Primary Outcome: Number of Participants Reporting Solicited Injection Site Reactogenicity Events
Description: Injection site AEs solicited on a memory aid provided to participants included Pain, Tenderness, Itching/Pruritus, Ecchymosis/Bruising (functional grade based on interference with daily activities), Ecchymosis/Bruising (any measured value >0mm), Erythema/Redness (functional grade), Erythema/ Redness (any measured value >0mm), Induration/Swelling (functional grade), and Induration/Swelling (any measured value >0mm). Participants are considered reporting the injection site AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The safety population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants | 11 | 35 | 5 | 16 | 11 | 38 | 3 | 14 | 12 | 30

6. Primary Outcome: Number of Participants Reporting Solicited Systemic Reactogenicity Events
Description: Systemic AEs solicited on a memory aid provided to participants included Elevated Oral Temperature, Feverishness, Fatigue, Malaise, Myalgia, Arthralgia, Headache, and Nausea. Participants are considered reporting the systemic AE if they reported mild or greater severity at any time during the 8 days at or following the first vaccination.
Time Frame: Day 1 through Day 8
Population: The safety population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants | 12 | 24 | 8 | 6 | 16 | 16 | 7 | 10 | 10 | 20

7. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater on Day 22 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: The modified intent-to-treat (mITT) population includes all participants who received at least one study vaccination and contributed both pre- and at least one post-study vaccination venous blood samples for HAI antibody assays for which valid results were reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 49 [31 to 66] | 88 [73 to 96] | 75 [53 to 90] | 89 [65 to 99] | 20 [9 to 36] | 59 [43 to 74] | 55 [32 to 77] | 94 [70 to 100] | 11 [2 to 28] | 9 [2 to 23]

8. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater on Day 22 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 69 [51 to 83] | 98 [87 to 100] | 92 [73 to 99] | 100 [81 to 100] | 43 [27 to 59] | 66 [50 to 80] | 75 [51 to 91] | 94 [70 to 100] | 4 [0 to 18] | 3 [0 to 15]

9. Primary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion on Day 22 Against the 2017 Influenza A/H7N9 Study Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after study vaccination is Day 22.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 49 [31 to 66] | 88 [73 to 96] | 75 [53 to 90] | 83 [59 to 96] | 20 [9 to 36] | 52 [37 to 68] | 55 [32 to 77] | 88 [62 to 98] | 7 [1 to 24] | 6 [1 to 19]

10. Primary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion on Day 22 Against the 2017 Influenza A/H7N9 Study Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after study vaccination is Day 22.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 69 [51 to 83] | 98 [87 to 100] | 83 [63 to 95] | 100 [81 to 100] | 43 [27 to 59] | 64 [48 to 78] | 75 [51 to 91] | 94 [70 to 100] | 4 [0 to 18] | 3 [0 to 15]

11. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies on Day 8 Against the 2017 Influenza A/ H7N9 Vaccine Virus
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 7 days post study vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 13.9 [9.3 to 20.7] | 54.2 [33.4 to 87.7] | 36.2 [21.3 to 61.3] | 113.9 [62.2 to 208.5] | 9.9 [7.0 to 14.0] | 18.1 [12.1 to 27.2] | 16.8 [9.2 to 30.8] | 91.8 [46.8 to 180.0] | 6.1 [4.6 to 8.1] | 6.1 [4.8 to 7.7]

12. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Hemagglutination Inhibition (HAI) Antibodies on Day 181 Against the 2017 Influenza A/ H7N9 Vaccine Virus
Description: Blood was collected for HAI assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 180 days post study vaccination (Day 181).
Time Frame: Day 181
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 27 | 34
titer | 10.5 [7.2 to 15.2] | 40.0 [25.6 to 62.4] | 35.1 [19.2 to 64.2] | 79.5 [40.6 to 155.6] | 9.9 [6.4 to 15.3] | 11.5 [8.3 to 15.9] | 9.5 [6.3 to 14.4] | 42.7 [23.3 to 78.1] | 5.1 [4.9 to 5.3] | 6.2 [4.8 to 7.9]

13. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neutralizing (Neut) Antibodies on Day 8 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 7 days post study vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 34.3 [21.4 to 55.1] | 153.2 [91.6 to 256.1] | 108.9 [62.4 to 189.8] | 482.5 [270.5 to 860.9] | 17.5 [12.1 to 25.2] | 31.4 [21.0 to 47.0] | 45.2 [20.8 to 97.9] | 320.0 [166.4 to 615.3] | 5.9 [4.8 to 7.3] | 7.0 [5.0 to 9.9]

14. Secondary Outcome: Geometric Mean Titers (GMT) of Serum Neutralizing (Neut) Antibodies on Day 181 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for Neutralizing assay which was conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 180 days post study vaccination (Day 181).
Time Frame: Day 181
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 19 | 16 | 27 | 34
titer | 24.1 [15.4 to 37.5] | 105.3 [65.8 to 168.2] | 73.4 [38.0 to 141.6] | 296.3 [147.4 to 595.6] | 14.3 [9.5 to 21.4] | 17.0 [12.2 to 23.9] | 34.6 [15.2 to 78.4] | 110.7 [56.1 to 218.4] | 5.4 [4.9 to 5.9] | 10.2 [7.8 to 13.4]

15. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Hemagglutination Inhibition (HAI) Antibodies on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for HAI assay which was conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 18.7 [12.2 to 28.5] | 92.7 [62.4 to 137.6] | 62.6 [35.3 to 111.0] | 166.3 [87.5 to 315.9] | 9.0 [6.5 to 12.6] | 21.0 [14.6 to 30.0] | 27.3 [14.5 to 51.4] | 146.7 [80.1 to 268.7] | 5.3 [4.8 to 5.9] | 6.1 [4.8 to 7.8]

16. Secondary Outcome: Geometric Mean Titers (GMTs) of Serum Neutralizing (Neut) Antibodies on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for Neutralizing assay which was conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The geometric mean titer was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
titer | 98.5 [59.8 to 162.2] | 515.4 [367.1 to 723.5] | 329.4 [192.5 to 563.6] | 1015.9 [785.2 to 1314.5] | 39.3 [23.6 to 65.5] | 102.1 [64.9 to 160.8] | 171.5 [82.6 to 356.0] | 744.8 [449.7 to 1233.5] | 7.0 [5.1 to 9.5] | 10.1 [7.2 to 14.1]

17. Secondary Outcome: Number of Participants Reporting Medically-Attended Adverse Events (MAAEs), New-Onset Chronic Medical Conditions (NOCMCs), and Potentially Immune-Mediated Medical Conditions (PIMMCs)
Description: Participants were queried at each visit for the occurrence of medically-attended adverse events (MAAEs), including new-onset chronic medical conditions (NOCMCs) and potentially immune-mediated medical conditions (PIMMCs) throughout the duration of the study.
Time Frame: Day 1 through Day 366
Population: The safety population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants
  MAAE | 5 | 8 | 5 | 6 | 13 | 7 | 8 | 4 | 10 | 3
  NOCMC | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
  PIMMC | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Number of Participants Reporting Unsolicited Non-serious AEs
Description: Adverse events were defined as any untoward medical occurrence in a participant administered a pharmaceutical product regardless of its causal relationship to the study treatment. Non-serious AEs were collected from participants at follow up visits through 21 days after study vaccination.
Time Frame: Day 1 through Day 22
Population: The safety population includes all participants who received study vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 38 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 29 | 35
Participants | 9 | 10 | 3 | 4 | 15 | 10 | 7 | 5 | 8 | 7

19. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater on Day 8 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm and stratum from the available results at 7 days post second vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 28 [14 to 45] | 65 [48 to 79] | 63 [41 to 81] | 83 [59 to 96] | 18 [7 to 33] | 41 [26 to 57] | 35 [15 to 59] | 81 [54 to 96] | 7 [1 to 24] | 6 [1 to 19]

20. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater on Day 181 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm and stratum from the available results at 180 days post second vaccination (Day 181).
Time Frame: Day 181
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 27 | 34
percentage of participants | 20 [8 to 37] | 55 [38 to 71] | 54 [33 to 74] | 78 [52 to 94] | 18 [7 to 33] | 25 [13 to 40] | 20 [6 to 44] | 56 [30 to 80] | 0 [0 to 13] | 6 [1 to 20]

21. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater on Day 8 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm and stratum from the available results at 7 days post study vaccination (Day 8).
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 53 [35 to 70] | 80 [64 to 91] | 79 [58 to 93] | 100 [81 to 100] | 33 [19 to 49] | 48 [32 to 63] | 55 [32 to 77] | 94 [70 to 100] | 4 [0 to 18] | 9 [2 to 23]

22. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater on Day 181 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm and stratum from the available results at 180 days post study vaccination (Day 181).
Time Frame: Day 181
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 19 | 16 | 27 | 34
percentage of participants | 31 [17 to 49] | 75 [59 to 87] | 67 [45 to 84] | 94 [73 to 100] | 23 [11 to 38] | 32 [19 to 48] | 42 [20 to 67] | 88 [62 to 98] | 0 [0 to 13] | 9 [2 to 24]

23. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion on Day 8 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 8 is 7 days post study vaccination.
Time Frame: Day 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 28 [14 to 45] | 60 [43 to 75] | 58 [37 to 78] | 83 [59 to 96] | 18 [7 to 33] | 34 [20 to 50] | 35 [15 to 59] | 75 [48 to 93] | 4 [0 to 18] | 3 [0 to 15]

24. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion on Day 181 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the HAI assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 181 is 180 days post study vaccination.
Time Frame: Day 181
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 27 | 34
percentage of participants | 20 [8 to 37] | 53 [36 to 68] | 50 [29 to 71] | 72 [47 to 90] | 18 [7 to 33] | 18 [8 to 33] | 20 [6 to 44] | 50 [25 to 75] | 0 [0 to 13] | 3 [0 to 15]

25. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion on Day 8 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 7 days after study vaccination is Day 8.
Time Frame: Day 8
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 36 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 53 [35 to 70] | 80 [64 to 91] | 75 [53 to 90] | 100 [81 to 100] | 33 [19 to 49] | 48 [32 to 63] | 55 [32 to 77] | 88 [62 to 98] | 4 [0 to 18] | 9 [2 to 23]

26. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion on Day 181 Against the 2017 Influenza A/H7N9 Vaccine Virus
Description: Blood was collected for the Neutralizing assay conducted with the 2017 H7N9 vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 180 days after study vaccination is Day 181.
Time Frame: Day 181
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 19 | 16 | 27 | 34
percentage of participants | 31 [17 to 49] | 73 [56 to 85] | 63 [41 to 81] | 94 [73 to 100] | 23 [11 to 38] | 32 [19 to 48] | 42 [20 to 67] | 88 [62 to 98] | 0 [0 to 13] | 9 [2 to 24]

27. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Titer of 1:40 or Greater on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for the HAI assay conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with HAI titer >= 1:40 was calculated for each study arm and stratum from the available results at 21 days post second vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 34 [19 to 52] | 85 [70 to 94] | 75 [53 to 90] | 94 [73 to 100] | 15 [6 to 30] | 45 [30 to 61] | 55 [32 to 77] | 94 [70 to 100] | 0 [0 to 12] | 3 [0 to 15]

28. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Titer of 1:40 or Greater on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for the Neutralizing assay conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. The percentage of participants with Neut titer >= 1:40 was calculated for each study arm and stratum from the available results at 21 days post study vaccination (Day 22).
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 74 [57 to 88] | 98 [87 to 100] | 96 [79 to 100] | 100 [81 to 100] | 50 [34 to 66] | 84 [70 to 93] | 90 [68 to 99] | 100 [79 to 100] | 4 [0 to 18] | 6 [1 to 19]

29. Secondary Outcome: Percentage of Participants Achieving Hemagglutination Inhibition (HAI) Antibody Seroconversion on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for the HAI assay conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as HAI pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. Day 22 is 21 days post study vaccination.
Time Frame: Day 22
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 34 [19 to 52] | 85 [70 to 94] | 75 [53 to 90] | 89 [65 to 99] | 15 [6 to 30] | 45 [30 to 61] | 55 [32 to 77] | 94 [70 to 100] | 0 [0 to 12] | 3 [0 to 15]

30. Secondary Outcome: Percentage of Participants Achieving Neutralizing (Neut) Antibody Seroconversion on Day 22 Against the 2013 Influenza A/H7N9 Vaccine Virus (Priming Vaccine Virus)
Description: Blood was collected for the Neutralizing assay conducted with the 2013 H7N9 priming vaccine virus as the antigen. Each sample was tested at least twice per the laboratory's standard operating procedure, and the geometric mean of the replicate results was calculated as that sample's result. Seroconversion was defined as Neut pre-vaccination titer <1:10 and post-vaccination titer >= 1:40 or pre-vaccination titer >= 1:10 and minimum 4-fold rise in post-vaccination antibody titer. 21 days after study vaccination is Day 22.
Time Frame: Day 22
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
Number analyzed (Participants) | 35 | 40 | 24 | 18 | 40 | 44 | 20 | 16 | 28 | 35
percentage of participants | 74 [57 to 88] | 98 [87 to 100] | 96 [79 to 100] | 100 [81 to 100] | 50 [34 to 66] | 84 [70 to 93] | 90 [68 to 99] | 100 [79 to 100] | 4 [0 to 18] | 3 [0 to 15]

ADVERSE EVENTS:
Time Frame: Solicited events and clinical safety laboratory AEs were collected from the time of study vaccination through 7 days after study vaccination. Unsolicited, non-serious AEs were collected from the time of study vaccination through approximately 21 days after study vaccination. SAEs, MAAEs, including NOCMCs and PIMMCs were collected from the time of study vaccination through approximately 12 months after study vaccination
Description: AEs were defined according to ICH E6. Any medical condition present at the time of screening was considered baseline and was not reported as an AE. If the severity of any pre-existing medical condition increased, it was recorded as an AE.
Arm/Group | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV|2017 A/H7N9 IIV | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 | A/H7 IIV Naïve |2017 A/H7N9 IIV | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40 | 0/24 | 0/18 | 0/40 | 0/44 | 0/20 | 0/16 | 0/29 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/40 | 0/24 | 0/18 | 0/40 | 0/44 | 0/20 | 0/16 | 1/29 | 0/35
Other Adverse Events (participants affected / at risk) | 25/38 | 37/40 | 12/24 | 16/18 | 29/40 | 40/44 | 13/20 | 15/16 | 19/29 | 34/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV (N=38) | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 (N=40) | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV (N=24) | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 (N=18) | 2013 A/H7N9 IIV|2017 A/H7N9 IIV (N=40) | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 (N=44) | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV (N=20) | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 (N=16) | A/H7 IIV Naïve |2017 A/H7N9 IIV (N=29) | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03 (N=35)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV (N=38) | 2013 A/H7N9 IIV+MF59|2017 A/H7N9 IIV+AS03 (N=40) | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV (N=24) | 2013 A/H7N9 IIV+AS03|2017 A/H7N9 IIV+AS03 (N=18) | 2013 A/H7N9 IIV|2017 A/H7N9 IIV (N=40) | 2013 A/H7N9 IIV|2017 A/H7N9 IIV+AS03 (N=44) | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV (N=20) | 2013 A/H7N9 IIV + MF59 or AS03 Then 2013 A/H7N9 IIV |2017 A/H7N9 IIV+AS03 (N=16) | A/H7 IIV Naïve |2017 A/H7N9 IIV (N=29) | A/H7 IIV Naïve |2017 A/H7N9 IIV+AS03 (N=35)
Ocular Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling of Eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 7 (7) | 15 (15) | 3 (3) | 2 (2) | 11 (11) | 9 (9) | 5 (5) | 6 (7) | 7 (7) | 10 (10)
Feeling Hot (General disorders) | 2 (2) | 4 (4) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 2 (2) | 1 (1) | 3 (3) | 5 (5)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Injection Site Erythema (General disorders) | 5 (5) | 10 (10) | 3 (3) | 4 (4) | 5 (5) | 10 (10) | 1 (1) | 5 (5) | 8 (8) | 7 (7)
Injection Site Haemorrhage (General disorders) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 0 (0) | 6 (6) | 0 (0) | 2 (2) | 1 (1) | 4 (4)
Injection Site Induration (General disorders) | 1 (1) | 7 (7) | 1 (1) | 4 (4) | 2 (2) | 7 (7) | 1 (1) | 3 (3) | 2 (2) | 8 (8)
Injection Site Pain (General disorders) | 0 (0) | 22 (22) | 0 (0) | 8 (9) | 2 (2) | 18 (18) | 1 (1) | 13 (13) | 3 (3) | 17 (17)
Injection Site Pain (Tenderness) (General disorders) | 7 (7) | 31 (31) | 1 (1) | 14 (14) | 6 (6) | 34 (34) | 1 (1) | 13 (13) | 4 (4) | 28 (28)
Injection Site Pruritus (General disorders) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Malaise (General disorders) | 4 (4) | 9 (9) | 3 (3) | 2 (2) | 8 (9) | 6 (6) | 2 (2) | 3 (3) | 3 (3) | 5 (5)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaccination Site Lymphadenopathy (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (2) | 0 (0) | 2 (2) | 4 (4) | 2 (3) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Chest Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 3 (5) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 1 (1)
Blood Creatinine Increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hemoglobin Decreased (Investigations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Platelet Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
White Blood Cell Count Decreased (Investigations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 4 (5) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 1 (1) | 4 (4)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 11 (11) | 0 (0) | 1 (1) | 1 (1) | 8 (8) | 5 (5) | 2 (2) | 4 (4) | 9 (9)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 8 (8) | 11 (11) | 6 (6) | 4 (4) | 11 (12) | 8 (8) | 2 (2) | 7 (7) | 6 (6) | 9 (9)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Menopausal Symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone Lesion Excision (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-12-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03738241/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT03738241/SAP_001.pdf